CLINICAL TRIAL: NCT07353164
Title: Comparison of Open Versus Laparoscopic High Ligation Varicocelectomy For The Treatment Of Varicocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Irfan Jamil, Principal Investigator, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LahoreGeneralH13
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Varicocele
Keywords: Varicocelectomy; High ligation; Open surgery; Laparoscopic surgery; Postoperative wound infection
MeSH Terms: conditions — Varicocele; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Open high ligation varicocelectomy) (Experimental): Open high ligation varicocelectomy
  Interventions: Procedure: Open high ligation varicocelectomy
- Group B (Laparoscopic high ligation varicocelectomy) (Active Comparator): Laparoscopic high ligation varicocelectomy
  Interventions: Procedure: Laparoscopic high ligation varicocelectomy

INTERVENTIONS:
Procedure: Open high ligation varicocelectomy — High ligation of the dilated testicular veins was performed by an open approach through a lower abdominal incision. The spermatic cord structures were approached extraperitoneally, the testicular vein was identified, separated from the artery after identification, and divided with ligatures. Wound closure was performed in layers with absorbable sutures and skin closure with silk sutures.
  Arms: Group A (Open high ligation varicocelectomy)
Procedure: Laparoscopic high ligation varicocelectomy — High ligation of the testicular vein was performed laparoscopically by inserting three ports. The testicular vessels were approached intraperitoneally, the testicular vein was identified, clipped, and divided. Wound closure was performed using absorbable suture material, with skin closure using silk sutures.
  Arms: Group B (Laparoscopic high ligation varicocelectomy)

SUMMARY:
Varicocele is a common condition in which veins around the testis become enlarged, and it may be associated with scrotal discomfort and reduced fertility. Surgical treatment aims to stop the backward flow of blood in these veins so that the testicular environment improves. This randomized controlled trial was conducted in the Department of Urology, PGMI, Lahore General Hospital, Lahore, over a six-month period.

Male patients aged 20 to 60 years with diagnosed varicocele and planned varicocelectomy under general anesthesia were enrolled after informed consent. Patients with recurrent varicocele, secondary varicocele, associated undescended testis, or a history of orchidopexy were excluded. Eligible participants were allocated into two groups using a lottery method. In Group A, high ligation was performed by the open method through a lower abdominal incision, with identification and ligation of the dilated testicular veins at a high level. In Group B, high ligation was performed laparoscopically using three small ports, with the testicular vein identified, clipped, and divided. Standard perioperative care was provided, including intravenous antibiotics and postoperative analgesia.

The study compared the two techniques in terms of mean operation time , length of hospital stay , and wound infection . The hypothesis was that a difference existed between open and laparoscopic high ligation varicocelectomy regarding operation time, hospital stay, and wound infection.

ELIGIBILITY:
Inclusion Criteria:

* Male patients age 20-60 years.
* Patients with varicocele.
* Planned to undergo varicocelectomy under general anesthesia.

Exclusion Criteria:

* Patients with recurrent varicocele.
* Secondary varicocele.
* Associated undescended testis or history of orchidopexy.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 100 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Mean operative time | During the surgery
  Operative time was measured in minutes from skin incision until completion of skin closure (stitching).

SECONDARY OUTCOMES:
Length of hospital stay | Up to 30 days post-surgery
  Hospital stay was measured in days from the day of surgery until discharge from the hospital.
Wound infection rate | 10 days after surgery
  Wound infection was assessed at 10 days after surgery with confirmation by positive pus culture when discharge was present.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Zeshan Aziz, Principal Investigator — Lahore General Hospital, Lahore
Locations (1):
- Lahore General Hospital, Lahore, Lahore, Punjab Province, Pakistan